CLINICAL TRIAL: NCT03527199
Title: Prospective Comparison of Pelvic CT or MRI Plus Bone Scanning With 99mTc-MDP Bone Scan and/or 18F-NaF PET/CT to 18F- Fluciclovine PET/CT in VA Prostate Cancer Patients With BCR.
Brief Title: Prostate Cancer Patients With Biochemical Recurrence
Status: Completed | Type: Observational
Sponsor: Medhat Osman (U.S. Federal Agency)
Collaborators: Blue Earth Diagnostics (Industry)
Responsible Party: Sponsor-Investigator, Medhat Osman, MD, PhD, Attending Physician at St. Louis VA Healthcare System, Saint Louis VA Medical Center
Organization: Saint Louis VA Medical Center (U.S. Federal Agency)
Other Study IDs: 1201372
Record Dates: First submitted 2018-05-04; First posted 2018-05-17 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Patients With Prostate Cancer
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Pelvic CT or MRI + MDP bone scan + or - 18F-NaF PET/CT(SOC) — Standard of care-Pelvic CT or MRI and MDP bone scan + or - 18F-NaF PET/CT

SUMMARY:
Evaluation of detection rate of 18F-Fluciclovine compared to current standard of care imaging techniques within 30 days of the standard of care imaging study and a 6 month phone follow-up

DETAILED DESCRIPTION:
When BCR is present, detection of recurrence as well as the location, distribution and number of metastatic sites would determine the choice of subsequent management. In the search of malignancy in patients with BCR, standard of care tests include Pelvic CT or MRI (to look for recurrence and/or pelvic nodal metastases) and a planar bone scan to look for skeletal metastases. However, standard of care testing has a low diagnostic yield of only 11% of patients for visualizing sites of disease (5). Thus, there is a clear need for better imaging approaches. 18F-Fluciclovine is a synthetic amino acid PET tracer approved by the Food and Drug Administration in June of 2016 for the detection of sites of recurrence in men with rising prostate-specific antigen levels after prior primary treatment of prostate cancer (6), based on its diagnostic performance (7,8). However, there is a gap in the literature regarding prospective studies evaluation of detection rate of 18F-Fluciclovine compared to current standard of care imaging techniques. Therefore, 18F-Fluciclovine has already been approved by the FDA and covered CMS and insurance companies but is yet to be included in the NCCN guidelines in the work up of PCa patients with BCR.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 and ≤89
2. History of Prostate Cancer which required surgical resection or radiation
3. Documented Biochemical recurrence defined as a positive PSA any time after the initial diagnosis of prostate cancer which at that time required surgical resection or radiation and then had a negative result to a post treatment PSA.
4. Patient undergoing standard of care work up pelvic CT or MRI, 99mTc-MDP bone scan, and F18 NaF PET/CT.

   -

Exclusion Criteria:

1. BCR with negative 99mTc-MDP bone scan but 18F-NaF PET/CT was not able to be done.

-

Ages: 18 Years to 89 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Study Population: Male subjects age 18-89
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
In the settings of BCR, detection rate of 18F- Fluciclovine will be compared to that of standard of care (SOC) (pelvic CT or MRI plus 99mTc-MDP bone scan). | 3-6months from acquiring Fluciclovine exam
  Detection rate of 18F- Fluciclovine PET/CT will be compared to current standard of care imaging with or without 18F-NaF PET/CT based on all available clinical follow up data including histological reference standard when biopsy of suspected lesion(s) is performed.

SECONDARY OUTCOMES:
In the settings of BCR with negative standard of care 99mTc-MDP bone scan, detection rate of 18F- Fluciclovine wiill be compared to that of standard of care pelvic CT or MRI plus 18F-NaF PET/CT. | 3-6months from acquiring Fluciclovine exam
  In the setting of PCa patients with BCR, documenting a higher detection rate for 18F- Fluciclovine PET/CT compared to current standard of care imaging modalities could result in future use of 18F- Fluciclovine PET/CT as a "one stop shop" for those patients.

CONTACTS AND LOCATIONS:
Overall Officials: Medhat M Osman, MD,PhD, Principal Investigator — St. Louis VA Helathcare System
Locations (1):
- John Cochran VA Medical Center St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No